CLINICAL TRIAL: NCT04690868
Title: A Randomized, Open Label, Multi Dose, Cross Over Design Clinical Study to Evaluate the Pharmacokinetic Pharmacodynamic Characteristics and Safety of AD-213-A and AD-2131 After Oral Administration in Healthy Adult Subjects
Brief Title: A Study to Compare PK, PD and Safety of the AD-213-A and AD-2131
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-213PK/PD
Record Dates: First submitted 2020-12-22; First posted 2020-12-31 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-11

CONDITIONS: Gastroesophagus Reflux Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1 (Experimental): Period 1 : Reference Drug(AD-2131) Period 2 : Test Drug(AD-213-A)
  Interventions: Drug: AD-213-A; Drug: AD-2131
- ARM 2 (Experimental): Period 1 : Test Drug(AD-213-A) Period 2 : Reference Drug(AD-2131)
  Interventions: Drug: AD-213-A; Drug: AD-2131

INTERVENTIONS:
Drug: AD-213-A — 1 tablet administered before the breakfast during 5 days
Drug: AD-2131 — 1 tablet administered before the breakfast during 5 days

SUMMARY:
A study to compare safety, pharmacokinetics and pharmacodynamics of AD-213-A to AD-2131 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over 19 years of age.
* Weight is more than 50kg and BMI is more than 18.0 kg/m^2 , no more than 27.0 kg/m^2.
* Subject who has been judged to be eligible for clinical laboratory tests and electrocardiogram tests such as serum tests, hematology tests, blood chemistry tests, and urinary tests conducted within four weeks prior to the administration of clinical trials.
* Subjects who has heard and fully understood the detailed description of this clinical trial and have willingness to sign of informed consent in writing.

Exclusion Criteria:

* A subject who has a history that can affect the absorption, distribution, metabolism, or excretion of a drug.
* As a result of laboratory tests, the following figures: ALT or AST or total bilirubin > 1.5 times upper limit of normal range.
* As a result of laboratory tests, the following figures: Creatinine clearance < 80mL/min.
* Subjects who judged ineligible by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
AUCtau | From Day 1 up to Day 17
  Evaluation PK after multiple dose
Integrated gastric acidity(%Decrease form baseline) | 4 times from Day -1 to Day 17
  Evaluation PD after multiple dose

SECONDARY OUTCOMES:
Cmax | Day 1
  Evaluation PK after single dose
AUClast | Day 1
  Evaluation PK after single dose
AUCinf | Day 1
  Evaluation PK after single dose
Tmax | Day 1
  Evaluation PK after single dose
t1/2 | Day 1
  Evaluation PK after single dose
CL/F | Day 1
  Evaluation PK after single dose
Vd/F | Day 1
  Evaluation PK after single dose
Cmax,ss | From Day 1 up to Day 17
  Evaluation PK after multiple dose
Cmin,ss | From Day 1 up to Day 17
  Evaluation PK after multiple dose
AUCinf | From Day 1 up to Day 17
  Evaluation PK after multiple dose
Tmax,ss | From Day 1 up to Day 17
  Evaluation PK after multiple dose
t1/2 | From Day 1 up to Day 17
  Evaluation PK after multiple dose
CLss/F | From Day 1 up to Day 17
  Evaluation PK after multiple dose
Vdss/F | From Day 1 up to Day 17
  Evaluation PK after multiple dose
Integrated gastric acidity(Variations form baseline) | 4 times from Day -1 to Day 17
  Evaluation PD after multiple dose
Percentage of time to maintain gastric pH 4.0 or higher | 4 times from Day -1 to Day 17
  Evaluation PD after multiple dose

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No